CLINICAL TRIAL: NCT05865678
Title: Musculoskeletal Health in Adult Haematoloigcal Cancer Survivors - a Mixed Methods Study
Brief Title: Musculoskeletal Health in Adult Haematological Cancer Survivors
Acronym: SKETCh
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: CFTsp167
Record Dates: First submitted 2023-04-24; First posted 2023-05-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Lymphoma; Leukemia; Cancer Survivors; Musculoskeletal Complication
MeSH Terms: conditions — Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (32):
- 5-10 years post cancer treatment; male; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; male; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; male; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; male; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; female; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; female; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; female; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 5-10 years post cancer treatment; female; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; male; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; male; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; male; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; male; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; female; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; female; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; female; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 11-20 years post cancer treatment; female; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; male; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; male; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; male; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; male; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; female; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; female; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; female; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 21-30 years post cancer treatment; female; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; male; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; male; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; male; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; male; age at diagnosis 70+
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; female; age at diagnosis 18-30
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; female; age at diagnosis 31-50
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; female; age at diagnosis 51-70
  Interventions: Other: Not an intervention study
- 30 years + post cancer treatment; female; age at diagnosis 70+
  Interventions: Other: Not an intervention study

INTERVENTIONS:
Other: Not an intervention study — This is a study administering questionnaire and interviews using mixed quantitative and qualitative methodology with the aim to describe and evaluate musculoskeletal health of adult haematological cancer survivors and its impact to survivors.

SUMMARY:
Haematological cancer treatment often includes use of high dose glucocorticoids (steroids), chemotherapy and radiotherapy and current evidence suggests that these patients may have lower bone mineral density after treatment when compared to the general population which can predispose them to increased risk of fragility fractures. Evidence of the impact of these musculoskeletal burden to patients (e.g. quality of life) are not available.

This study aims to describe musculoskeletal complications experienced by long-term haematological cancer survivors and examine the impact of the burden from the patient perspective. The study will be conducted in 2 parts; a questionnaire study and an interview study to help understand the extent of musculoskeletal problems experienced by this group of patients and the impact of this on quality of life.

ELIGIBILITY:
Questionnaire study

Inclusion Criteria:

1. Age 18 or above at diagnosis of haematological cancer
2. Diagnosis of haematological cancers: lymphoma or leukaemia
3. Cancer survivors as recorded in the local database of lymphoma and haematopoietic stem cell transplant database
4. Able to give written informed consent
5. Able to read and understand English

Exclusion Criteria:

1.Currently receiving any active cancer treatment

Interview study

Inclusion Criteria:

1. Age 18 or above at diagnosis of haematological cancer
2. Diagnosis of haematological cancers: lymphoma or leukaemia
3. Cancer survivors as recorded in the local database of lymphoma and haematopoietic stem cell transplant database
4. Able to give written or verbal informed consent
5. Able to read and understand English

Exclusion Criteria:

1 .Currently receiving any active cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from The Christie NHS Foundation Trust local haematology and lymphoma survivors' clinical patient databases. The haematology database used is the HSCT database that records all haematology patients that have undergo haematopoietic stem cell transplant. For lymphoma patients, the ADAPT (Managed Local Follow up of Long-Term Lymphoma Survivors) database will be used which records lymphoma patients that are cured and had 5 years regular hospital follow up post treatment.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Questionniare study: To measure prevalence of musculoskeletal conditions and related symptoms experienced by adult lymphoma and leukaemia survivors | overall length of the study - 6 months
  Musculoskeletal conditions and related symptoms will be recorded by patients on the study specific questionnaire and the validated questionnaire Nordic musculoskeletal questionnaire (NMQ-E) and gait, arms, legs and spine (GALS) assessment
Questionniare study: To calculate the 10-year probability of hip fracture and major osteoporotic fracture (clinical spine, forearm, hip or shoulder fracture) of adult lymphoma and leukaemia survivors | overall length of the study - 6 months
  The 10-year probability of hip fracture and major osteoporotic fracture (clinical spine, forearm, hip or shoulder fracture) of adult lymphoma and leukaemia survivors will be calculated using the Fracture Risk Assessment Tool (FRAX) and Q-Fracture calculator.
Questionniare study: To measure prevalence of sarcopenia and frailty among adult lymphoma and leukaemia survivors | overall length of the study - 6 months
  Validated questionniares will be used to assess if patients have sarcopenia (SARC-F questionnaire) and frailty (FiND questionnaire).
Questionniare study: To assess quality of life and musculoskeletal function related quality of life of adult lymphoma and leukaemia survivors | overall length of the study - 6 months
  This will be assessed using validated questionnaires - Short Form Survey (SF36) and Short Musculoskeletal Function Assessment (SMFA).
Interivew study: To describe experience of adult lymphoma and leukaemia survivors on musculoskeletal health, musculoskeletal related care and musculoskeletal health information provision. | overall length of the study - 6 months
  Semi-structured qualitative interviews will be conducted with a topic guide to ensure same broad topics are explored in the interviews on musculoskeletal health experience, care and information provision.

SECONDARY OUTCOMES:
Questionnaire study: To describe the likely risk factors that may be associated with musculoskeletal consequences of adult lymphoma and leukaemia survivors Impact of musculoskeletal health | overall length of the study - 6 months
  This will be assessed using regression analysis to determine risk factors that may be associated with poor musculoskeletal health

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No